CLINICAL TRIAL: NCT04194268
Title: Pancreatic Cancer and Carbon Ion Radiotherapy
Acronym: PACK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Head of Department, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RADONK-PACK-2019
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional arm (Experimental): Carbon Ion Radiation 12 x 4 Gy (RBE) within 2 weeks
  Interventions: Radiation: Carbon Ion

INTERVENTIONS:
Radiation: Carbon Ion — 12 x 4 Gy (RBE)

SUMMARY:
Irradiation of non-operable pancreatic cancer with carbon ions (C12). This therapy is expected to be more effective than the current Gold Standard of photon irradiation applied in the case of non-operable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, inoperable primary or local recurrent pancreatic cancer
* Written informed consent (must be available before enrollment in the trial)
* Karnofsky performance score > 60 or ECOG-status 0/1 (at least: patient should be able to take care of himself, although daily-life activity or work is not possible)
* Age ≥ 18 years

Exclusion Criteria:

* No clear difference between tumor edge and upper gastrointestinal tract in baseline imaging
* Extensive lymphatic metastases
* Disability of subject to understand character and individual consequences of the clinical trial
* Distant metastases
* Previous radiotherapy of the upper abdomen
* Active medical implants (e.g. pacemaker, defibrillator), contradicting radiotherapy at HIT
* Participation in another clinical study or observation period of competing trials, respectively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2025-10-09 (Estimated); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
survival | 12 month after radiation
  overall survival

SECONDARY OUTCOMES:
toxicity outcomes | 48 Month after radiatoin
  Incidence of grade 3/4 NCI-CTC-AE toxicity
survival | 12 month after radiation
  Progression free survival
Blood Parameters Ca 19-9 | 48 Month after radiation
  Change in Ca 19-9
Blood Parameters CEA | 48 Month after radiation
  Change in CEA levels
Quality of life (QLQ) EORTC QLQ C30 | 48 Month after radiation
  Change on scoring on EORTC QLQ C30
Quality of life EORTC QLQ Pan26 | 48 Month after radiation
  Change on scoring EORTC QLQ Pan26

CONTACTS AND LOCATIONS:
Locations (1):
- University Hopsital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Liermann J, Naumann P, Hommertgen A, Pohl M, Kieser M, Debus J, Herfarth K. Carbon ion radiotherapy as definitive treatment in non-metastasized pancreatic cancer: study protocol of the prospective phase II PACK-study. BMC Cancer. 2020 Oct 1;20(1):947. doi: 10.1186/s12885-020-07434-8. PMID 33004046